CLINICAL TRIAL: NCT06564675
Title: Accuracy of EEG Slow Wave Activity in Predicting Favourable Outcome in Patients With Hypoxic Brain Injury - A Substudy of STEPCARE Trial
Acronym: PROPEASTEPCARE
Status: Recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: University of Oulu (Other); Skane University Hospital (Other); Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Tampere University (Other); Charite University, Berlin, Germany (Other); Oslo University Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Johanna Hastbacka, associate professor, Tampere University
Other Study IDs: STEPCARE-EEG
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA patients: OHCA patients, randomized to STEPCARE Trial. The patients are recruiten to this substudy in selected centers with access to the Brainstatus device for recording of cEEG.
  Adult patients who remain comatose after sustained ROSC after OHCA are eligible to the STEPCARE Trial. Exclusion criteria are pregnancy, previous randomization to STEPCARE, trauma or hemorrhage as reasons for arrest, suspected or confirmed intracranial hemorrhage, and specifically for this study allergy to adhesive material and injured skin in the frontal-temporal area, that prevents adhesion of the Brainstatus electrode.
  Interventions: Diagnostic Test: C-Trend Index

INTERVENTIONS:
Diagnostic Test: C-Trend Index — C-trend-Index is collected blinded from the patients using Brainstatus device. The device shows and collects also cEEG. These are analyzed retrospectively after all study patients have their 6-month follow-up data collected. The intervention does not affect clinical management or decision-making.
  Other Names: visual assessment of cEEG

SUMMARY:
This is an observational substudy embedded in the STEPCARE Trial. The study involves EEG analysis, covered by the ethics approval of STEPCARE Trial. The investigators aim to compare the accuracy of a continuously measured algorithm-based EEG index, C-Trend Index, with retrospective visual analysis of continuous EEG in predicting favorable functional outcome in adult patients treated in intensive care units after out-of-hospital cardiac arrest. The primary hypothesis is that the accuracy of C-Trend Index has at least 10% better accuracy in predicting favorable outcome than the visual analysis of cEEG, when assessed early, 9-12 hours after return of spontaneous circulation (ROSC).

DETAILED DESCRIPTION:
STEPCARE Trial (Clinical trials identifier:NCT05564754) includes adult out-of-hospital cardiac arrest (OHCA) patients, with sustained ROSC, who remain comatose after resuscitation. STEPCARE is a factorial Trial, where all participants are randomized regarding three different interventions (minimal or deep sedation, target mean arterial pressure 65mmHg or 85mmHg, temperature management with or without a device). Patients with suspected or confirmed intracerebral hemorrhage, trauma or hemorrhage as reasons of arrest, those previously randomized to STEPCARE and patients with allergy to adhesive material or skin injury in the frontal-temporal area will be excluded (the latter two specific to this substudy).

The investigators aim to assess whether a new, algorithm-based index derived from continuous EEG (cEEG) recording is superior to retrospective visual analysis of cEEG in predicting functional outcome after OHCA, assessed restrospectively from early phase recordings, using the best hour within the 9-12-hour time interval after ROSC.

The cEEG will be collected using a commercially available Brainstatus device in selected centers participating in the STEPCARE Trial. cEEG will be visible to clinical team in centers using cEEG in routine monitoring, but blinded for those who do not routinely monitor cEEG in OHCA patients. C-Trend Index is blinded to clinicians and researchers, and will be analyzed retrospectively, after the primary outcome has been collected of the last patient of this substudy.

The primary outcome of this substudy is the functional outcome 6 months after OHCA, defined as modified Rankin Scale score (dichotomized as favourable mRS 0-3, and unfavourable mRS 4-6), assessed by blinded outcome assessors.

The investigators will compare accuracy (with separate comparisons of sensitivity and specificity) of C-Trend Index 9-12 hours after ROSC with the visual assessment of cEEG. C-Trend Index above a predefined cut-off value 20 is defined as indicative of favorable outcome, while in the visual assessment continuous or nearly continuous normal-voltage background without abundant discharges is considered indicative of favorable outcome .

To demonstrate a 10% difference in the accuracy, a sample size of 271 patients is needed. To account for loss of patients due to early wake-up, loss of follow-up, and technical issues in recordings the investigators aim at recruiting 300 patients.

As secondary research questions the study will also assess:

* The predictive accuracy off C-Trend Index in predicting unfavorable functional outcome, compared with visual analysis of cEEG
* The predictive accuracy of C-Trend Index using cut-off values 50 and 80 at 9-12 hours from ROSC in predicting favorable and unfavorable functional outcome
* Whether the predictive ability or the optimal cut-off value of C-Trend Index in predicting favorable and unfavorable functional outcome is affected by the three different interventions of the STEPCARE study

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* OHCA, with sustained ROSC
* Unconscious after ROSC
* No limitations to full life support
* Randomized to STEPCARE Trial in a participating center with Brainstatus device available

Exclusion Criteria:

* age <18
* Previously randomized to STEPCARE
* Trauma or hemorrhage as the reasons for arrest
* Suspected or confirmed intracerebral hemorrhage
* Allergy to adhesive material
* Damaged skin at the frontal-temporal are preventing electrode attachment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients resuscitated from OHCA
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Predictive accuracy of C-Trend Index >20 for favorable functional outcome | cEEG is recorded at least 24 hours after inclusion to the study, or until the patient awakens to respond to verbal commands. Data collected from recorded cEEG and C-Trend Index are assessed from the time point of 9-12 hours from ROSC.
  Predictive accuracy of C-Trend Index >20 at 9-12 hours from ROSC compared to retrospective visual analysis of cEEG in predicting favourable functional outcome defined as modified Rankin Scale 0-3 six months after OHCA

SECONDARY OUTCOMES:
Predictive accuracy of C-Trend Index for unfavorable functional outcome | cEEG is recorded at least 24 hours after inclusion to the study, or until the patient awakens to respond to verbal commands. Data collected from recorded cEEG and C-Trend Index are assessed from the time point of 9-12 hours from ROSC.
  Predictive accuracy of C-Trend Index >20 at 9-12 hours from ROSC compared to retrospective visual analysis of cEEG in predicting unfavorable functional outcome defined as modified Rankin Scale 4-6 six months after OHCA
Predictive accuracy of C-Trend Index >50 and >80 for favorable functional outcome | cEEG is recorded at least 24 hours after inclusion to the study, or until the patient awakens to respond to verbal commands. Data collected from recorded cEEG and C-Trend Index are assessed from the time point of 9-12 hours from ROSC.
  Predictive accuracy of C-Trend Index >50 and >80 at 9-12 hours from ROSC compared to retrospective visual analysis of cEEG in predicting favorable functional outcome defined as modified Rankin Scale 4-6 six months after OHCA
Predictive accuracy of C-Trend Index >50 and >80 for unfavorable functional outcome | cEEG is recorded at least 24 hours after inclusion to the study, or until the patient awakens to respond to verbal commands. Data collected from recorded cEEG and C-Trend Index are assessed from the time point of 9-12 hours from ROSC.
  Predictive accuracy of C-Trend Index >50 and >80 at 9-12 hours from ROSC compared to retrospective visual analysis of cEEG in predicting unfavorable functional outcome defined as modified Rankin Scale 4-6 six months after OHCA
Do the interventions in the STEPCARE Trial affect the predictive accuracy of C-trend Index | cEEG is recorded at least 24 hours after inclusion to the study, or until the patient awakens to respond to verbal commands. Data collected from recorded cEEG and C-Trend Index are assessed from the time point of 9-12 hours from ROSC.
  Is the predictive ability or the optimal cut-off values of C-Trend Index in predicting favourable and unfavourable outcomes affected by the three different interventions of the STEPCARE study

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Kortelainen, MD, PhD, Study Director — University of Oulu
Locations (4):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hastbacka J, Westhall E, Moseby-Knappe M, Tiainen M, Lybeck A, Reinikainen M, Levin H, Skrifvars MB, Tirkkonen J, Jakobsen JC, Nielsen N, Toppila J, Admiraal MM, Kortelainen J. Accuracy of EEG Slow Wave Activity in Predicting Favorable Outcome in Patients With Hypoxic Brain Injury-A Protocol for a Substudy of the STEPCARE Trial. Acta Anaesthesiol Scand. 2025 Oct;69(9):e70126. doi: 10.1111/aas.70126. PMID 40958738